CLINICAL TRIAL: NCT00004036
Title: Phase I Trial of High Dose Chemotherapy Using Amifostine for In-Vivo Protection of GM-CSF Primed Progenitor Cells
Brief Title: Combination Chemotherapy Plus Amifostine in Treating Patients With Advanced Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Cleveland Clinic (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000066347; CCF-IRB-1907; IMMUNEX-001.G9701; NCI-V98-1424
Record Dates: First submitted 1999-12-10; First posted 2004-09-13 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Myeloproliferative Disorders; Drug/Agent Toxicity by Tissue/Organ; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; drug/agent toxicity by tissue/organ; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Drug-Related Side Effects and Adverse Reactions; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — sargramostim; Amifostine; Carboplatin; Cyclophosphamide

INTERVENTIONS:
Biological: sargramostim
Drug: amifostine trihydrate
Drug: carboplatin
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumors from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of amifostine plus combination chemotherapy in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effects of priming on the granulocyte and thrombocyte nadirs produced by high dose cyclophosphamide and carboplatin in patients with advanced malignancies. II. Determine the effects of amifostine on the granulocyte and thrombocyte nadirs produced by this same regimen when administered with sargramostim primed progenitor cells. III. Determine the maximum tolerated dose of cyclophosphamide and carboplatin that can be administered with sargramostim primed progenitor cells.

OUTLINE: This is a dose escalation study. Patients receive intravenous amifostine over 10 minutes on day 0, followed by intravenous cyclophosphamide and carboplatin consecutively over 5-15 minutes. Sargramostim is administered subcutaneously on days -7 to -2 and again beginning on day 1 until absolute neutrophil count is appropriate. Course is repeated every 28 days until disease progression or unacceptable toxic effects are observed. Nonresponding patients discontinue treatment after 2 courses. Patients are treated for a maximum of 6 courses. Groups of 3-6 patients receive escalating doses of cyclophosphamide and carboplatin until the maximum tolerated dose (MTD) is determined. If dose limiting toxicity (DLT) occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and the next lower dose is declared the MTD.

PROJECTED ACCRUAL: Approximately 24-30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced malignancies that are sensitive to cyclophosphamide/carboplatin therapy OR refractory to standard therapy, including, but not limited to: Ovarian epithelial cancer Colorectal cancer Breast cancer Sarcoma Non-small cell lung cancer Malignant melanoma Upper gastrointestinal cancers Small cell lung cancer

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 SWOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.5 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min OR Iothalamate clearance at least 60 mL/min Cardiovascular: No significant coronary artery disease (angina of New York Heart Association class 3 or greater) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No psychosis

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No more than 1 prior chemotherapy regimen for advanced or recurrent malignancies (not including adjuvant chemotherapy) No prior nitrosoureas or intravenous mitomycin No concurrent cytotoxic chemotherapy Endocrine therapy: At least 1 week since prior hormone therapy and recovered Concurrent corticosteroid therapy allowed Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Radiotherapy allowed to no more than 1 site in the thoracic or lumbar spine or pelvis Concurrent radiotherapy to a symptomatic lesion allowed after the first course of study treatment Surgery: At least 3 weeks since prior surgery and recovered (excluding recent biopsy or placement of an intravenous access device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: George Thomas Budd, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Cancer Center, Cleveland, Ohio, United States